CLINICAL TRIAL: NCT03379818
Title: Shape Bias Training as a Vocabulary Intervention for Late Talkers
Brief Title: Vocabulary Intervention for Late Talkers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to closures related to the Covid-19 pandemic.
Sponsor: University of Birmingham (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Andrea Krott, Dr, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG_17-142
Record Dates: First submitted 2017-12-06; First posted 2017-12-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Language Delay; Language Development Disorders
Keywords: Shape bias; Late Talkers
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Over a series of 9 weekly sessions, children diagnosed as Late Talkers will be assessed in different tasks that can be divided into 5 phases: Vocabulary and developmental assessments, initial cognitive assessments, training sessions, word learning test 1, and word learning test 2. Each group (shape training group and specific word training group) will receive a different training programme, however the other assessments will be identical across the groups. In the shape training group, participants will be taught to attend to shape when learning and extending novel labels. In the specific word training group, participants will be taught specific words that they do not know. Before and after the intervention, participants vocabulary will be assessed to compare which intervention enhances word learning. One year later, all participants will be assessed with a language test and a cognitive test. The same assessments will be used in both groups.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two possible groups. In both groups, they will receive an intervention, however participants and their parents will not know which one. At the end of the study, participants and their parents will be informed about which group they were in and a document containing a detailed description of each intervention will be provided to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific word training intervention (Experimental): This training programme will be similar to a typical word learning intervention. Infants will be introduced to 28 real objects and their names (e.g. biscuit, trousers). These objects will be divided into 7 sets of four words, and during each session, infants will be presented with one of this sets. Each session will consist of a 15 min play session in which each object will be presented at least 10 times and each object name will be mentioned at least 10 times. Additionally, techniques such as focused stimulation and modelling target words, which have proved to be useful for word learning, will be used.
  Interventions: Behavioral: Specific word training
- Shape training intervention (Experimental): In the shape training intervention, infants will be presented with four novel words paired with four novel sets of objects. Each set consists of two exemplars with the same shape but with different colors and textures, and a contrasting object. Each set will be presented in a play session, and the name of the objects will be mentioned at least 10 times. The other three sets of exemplars will be presented in the same way. Each session will last 15 minutes. This intervention is based on a study conducted by Smith and colleagues (2002), where they found that typically developing infants that are taught to attend to shape at 17 months old, can enhance significantly their word learning.
  Interventions: Behavioral: Shape training intervention

INTERVENTIONS:
Behavioral: Shape training intervention — This intervention is based on on a study conducted by Smith and colleagues (2002), where they found that teaching typically developing infants to attend to shape by the end of the second year of life significantly enhances their word learning. Participants will be taught that the significant property they should focus in when learning and extending novel labels is shape. This will be done through play-like sessions.
  Arms: Shape training intervention
Behavioral: Specific word training — In this intervention, participants will be taught the names of 28 real objects. The target words have been selected from the "Wordbank database", which is an open database that lists the proportion of children that know a specific word at a specific age. Twenty-eight words that are understood by 80% of the total child population at 25 months were randomly selected as target words. Techniques such as focused stimulation and modelling target words, which have proved to be useful for word learning, will be used.
  Arms: Specific word training intervention

SUMMARY:
Most studies regarding word learning have focused on understanding when and how infants learn words. At 24 months, typically developing infants know between 200 and 300 words and add new words to their vocabularies at a rapid rate. It is also during the first years of life that some principles that promote vocabulary learning are developed. The shape bias, which is a tendency to infer that objects that share the same shape will also share the same name, is the one that has been studied the most. At 24 months, typically developing infants use this principle as a strategy to learn novel words. In contrast, Late Talkers (children with a language delay in the absence of a physiological, cognitive or genetic disorder that may account for this delay) do not exhibit this preference. It has been found that teaching typically developing infants a shape bias prior to the end of the second year of life can boosts their word learning. Despite this, the possibility of teaching Late Talkers this principle and its effect on their vocabulary and language development has not been explored.

Over a series of 9 weekly sessions, Late Talkers (diagnosed by Language Therapists from the Birmingham Community Healthcare National Health Services Foundation Trust, United Kingdom) will be introduced to one of two possible interventions: a shape bias intervention and a more conventional intervention called "specific word intervention". Both interventions will be compared after 9 weeks. One year later, a follow up study will be conducted to assess the long-term effects each intervention has in word learning. Participants will be referred by a Speech and Language Therapists from the Birmingham Community Healthcare National Health Services Foundation Trust, United Kingdom, and all assessments and interventions will take place at the Infant and Child Lab at the University of Birmingham, United Kingdom.

DETAILED DESCRIPTION:
The objectives of the present study are:

A. To investigate whether it is possible to teach Late Talkers to attend to objects' shapes as a useful property for learning and generalizing novel object labels.

B. To assess the benefits that this intervention programme has on Late Talkers' short-term vocabulary development compared to an intervention where infants will be taught specific words ('specific word' intervention).

C. Assess whether the success of teaching Late Talkers a shape bias for noun extension is related to their sensitivity to object shape similarities.

D. Assess whether the success of teaching Late Talkers a shape bias for noun extension is related to their ability of sustain their attention to novel objects that are presented to them.

E. To assess the benefits of the intervention programme on language and cognitive development one year after the intervention compared to the 'specific word' intervention

ELIGIBILITY:
Inclusion Criteria:

* Children (boys and girls) between 24 and 48 months.
* Children from Birmingham (United Kingdom) and its surrounding areas.
* Monolingual English native speakers
* Children with a moderate or severe language delay, as diagnosed by a Speech and Language Therapist of the Birmingham Community Healthcare National Health Service Foundation Trust, United Kingdom.

Exclusion Criteria:

* Children with a developmental, physiological, neurological or cognitive disorder that could explain their language delay.
* Children with a mild language delay, as diagnosed by a Speech and Language Therapist of the Birmingham Community Healthcare National Health Service Foundation Trust, United Kingdom.
* Children that speak or know another language different than English, either as first or additional language.

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Krott, Dr, Study Director — University of Birmingham; Claudia Zuniga-Montanez, Principal Investigator — University of Birmingham
Locations (1):
- Infant and Child Laboratory, University of Birmingham, Edgbaston, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants recruited differs from the one described in the protocol as this study had to be stopped due to the covid-19 pandemic.
Groups:
- Specific Word Training Intervention: This training programme was similar to a typical word learning intervention and was the control group. Children were introduced to 28 real objects and their names (e.g. biscuit, trousers). These objects will be divided into 7 sets of four words, and during each session, children were presented with one of these sets. Each session consisted of a 15 min play session in which each object was presented at least 10 times and each object name mentioned at least 10 times. Additionally, techniques such as focused stimulation and modelling target words, which have proved to be useful for word learning, were used.
- Shape Training Intervention: In the shape training intervention, children were presented with four novel words paired with four novel sets of objects. Each set consisted of two exemplars with the same shape but with different colors and textures, and a contrasting object. Each set was presented in a play session, and the name of the objects were mentioned at least 10 times. The other three sets of exemplars were presented in the same way. Each session lasted 15 minutes. This intervention was based on a study conducted by Smith and colleagues (2002), where they found that typically developing infants that are taught to attend to shape at 17 months old, can enhance significantly their word learning.
Period: Overall Study
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Started | 12 | 14
Completed | 7 | 7
Not Completed | 5 | 7
Not completed — Closures due to the Covid-19 pandemic | 2 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Diagnosis or suspected diagnosis of Autism spectrum disorder (ASD) | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Specific Word Training Intervention | Shape Training Intervention | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the start of the study.
  Years | 2.61 (0.42) | 2.76 (0.52) | 2.69 (0.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Age of first words [Mean (Standard Deviation); unit: months] — Population: Two participants in each group were not yet using words to communicate at the beginning of the study as reported by parents.
  months
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 22.16 (3.25) | 21.25 (9.21) | 21.8 (6.23)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Shape Choices in Two Noun Extension Tests.
Description: Assessed using two noun extension tests with known and novel names and objects. The objective was to assess if participants would extend known or novel names to objects sharing the same shape. The test with known names was conducted in week 8. The test with novel names was conducted at week 9 after starting the intervention.
  In each test, participants completed 8 trials. For each trial, participants were shown an object and heard its name. They were then asked to get another object that was also called the same from a set of 3 objects shown to them (one object shared the same shape, a second one shared the same colour and a third one shared the same texture). The same procedure was used on each trial but the objects and names used were different each time.
  If participants learned a shape bias, they should have mainly chosen the objects that shared the same shape. Below we show the average percentage of shape choices in each group for both tests.
Time Frame: At week 8 after starting the interventions for known names and objects. At week 9 after starting the interventions for novel names and objects.
Measure: Mean (Standard Deviation); unit: percentage of shape choices
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 7 | 7
percentage of shape choices
  Known objects (week 8 after starting the intervention) | 37.50 (10.20) | 56.63 (18.37)
  Novel objects (week 9 after starting the intervention) | 34.69 (18.97) | 39.28 (13.36)

2. Primary Outcome: Assessment of Number of Words Known Before and After the Interventions.
Description: In order to assess the benefits of each intervention programme, parents/guardians filled in a vocabulary checklist before (week 1) and after (week 9) the interventions. We compared the vocabulary growth (receptive and expressive vocabulary) in the group of children that took part in the shape bias intervention programme with that of the group of children that took part in the 'specific word' intervention.
Time Frame: Parents/guardians filled in a vocabulary checklist before (week 1) and after (week 9) the interventions.
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 7 | 7
number of words
  Receptive (week 1 - vocabulary at the start of the study) | 207 (95.96) | 288.43 (87.11)
  Receptive (week 9 - vocabulary at the end of the study) | 263.86 (107.19) | 355.29 (106.81)
  Expressive (week 1 - vocabulary at the start of the study) | 62 (46.04) | 76.86 (83.77)
  Expressive (week 9 - vocabulary at the end of the study) | 146.86 (109.90) | 149.14 (151.35)

3. Primary Outcome: Long-term Effects of Each Intervention on Language Development.
Description: This was expected to be assessed with a language test. Due to closures related to the covid-19 pandemic, this assessment was not able to be conducted and the study was stopped.
Time Frame: Was expected to be assessed one year after the end of the intervention programme.
Population: Due to closures related to the covid-19 pandemic, this assessment was not able to be conducted and the study was stopped.
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Long-term Effects of Each Intervention on Visual Spatial Skills.
Description: Each child was expected to be assessed with a standardized visual spatial test. Due to closures related to the covid-19 pandemic, this assessment was not able to be conducted and the study was stopped.
Time Frame: Visual spatial skills assessed one year after the end of the intervention programme.
Population: as for outcome 3
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Long-term Effects of Each Intervention on Working Memory.
Description: Each child was expected to be assessed with a memory test. Due to closures related to the covid-19 pandemic, this assessment was not able to be conducted.
Time Frame: Was expected to be assessed one year after the end of the intervention programme.
Population: Due to closures related to the covid-19 pandemic, this assessment was not able to be conducted.
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Children's Sensitivity Towards Shape Similarities.
Description: Assessed by relating children's ability to sort objects by shape before the intervention.
Time Frame: Assessed in the first week of the intervention.
Measure: Mean (Standard Deviation); unit: percentage correctly sorted by shape
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 7 | 7
percentage correctly sorted by shape | 41.66 (19.83) | 42.85 (10.12)

7. Secondary Outcome: Children's Attention to Novel Objects.
Description: Assessed by relating children's sustained attention during the presentation of a video showing a person presenting and moving novel objects before the intervention.
  Note that two participants preferred not to complete this assessment, therefore they are not included in this analysis.
Time Frame: Assessed with an attention task in the first week of the intervention.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
Number analyzed (Participants) | 7 | 5
seconds
  Video 1 | 21.57 (10.71) | 14.45 (12.46)
  Video 5 | 4.16 (10.20) | 4.38 (9.79)

ADVERSE EVENTS:
Time Frame: This study was a language intervention where children played with toys and were then assessed to see what they learned, therefore no adverse effects were expected/monitored.
Description: This study was a language intervention where children played with toys and were then assessed to see what they learned. All objects used were similar to objects/toys children would encounter and play with in their everyday life. Additionally, parents/carers were present in the room at all times with the researcher and the participant. Due to the nature of the intervention, no adverse effects were expected, therefore no adverse effects were monitored/assessed.
Arm/Group | Specific Word Training Intervention | Shape Training Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The current project was stopped due to the Covid-19 pandemic. The follow-up was not able to be conducted due to closures, lockdowns and restrictions related to the Covid-19 pandemic. The number of participants was also smaller than planned due to the same reasons. Note that only a few participants were recruited through Birmingham Community Healthcare NHS Foundation Trust and others were recruited through community or social groups, or Language Through Play groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03379818/Prot_SAP_000.pdf